CLINICAL TRIAL: NCT06014112
Title: Predictive Value of Glycemic Parameters Measured With the Freestyle Libre Pro iQ During Acute Coronary Syndrome
Brief Title: Predictive Value of Glycemic Parameters Measured With the FSL Pro iQ During ACS
Acronym: FREESCA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RECHMPL22_0395
Record Dates: First submitted 2023-08-22; First posted 2023-08-28 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Acute Coronary Syndrome; Continuous Glucose Measurement; Glycemic Variability; Cardiovascular Event
Keywords: acute coronary syndrome; continuous glucose measurement; glycemic variability; cardiovascular event
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Freestyle Libre PRO iQ sensor (Experimental): Eligible patients
  Interventions: Device: Freestyle Libre Pro iQ

INTERVENTIONS:
Device: Freestyle Libre Pro iQ — Freestyle Libre Pro iQ is a professional sensor, marketed by the Abbott laboratory, for continuous, non-invasive interstitial glucose measurement allowing the recording of glycemic parameters for 2 weeks.
  The study will be offered to any subject with an ACS. The installation of the Freestyle Libre Pro iQ sensor will be performed upon admission to intensive care Cardiology and left in place for the duration of hospitalization. In case of the Freestyle Libre Pro iQ sensor defective or removed before discharge from hospital, and if the patient tolerates it, a new the Freestyle Libre Pro iQ sensor will be placed. If the duration of hospitalization exceeds 14 days, a 2nd sensor will be placed.

SUMMARY:
Disorders of glycemic regulation are common in patients hospitalized for acute coronary syndrome (ACS). Abnormal glycaemia is observed in 50% of cases, in 30-40% diabetes, and in 25-35% fasting hyperglycaemia or glucose intolerance.

Hyperglycemia is a major prognostic factor in ACS, with admission hyperglycemia having independent prognostic value for both short- and long-term major cardiovascular events (MACE), regardless of the presence of diabetes.

Metabolically, several situations can be distinguished:

* Hyperglycaemia occurs in known non-diabetic ACS subjects. It can be indicative of (i) Type 2 Diabetes or (ii) stress hyperglycaemia (diagnostic threshold for blood sugar varies according to learned societies, with HbA1c < 6.5%).
* Hyperglycaemia occurs in known diabetic ACS subjects Most studies use admission blood sugar as a predictor. However, it has recently been shown that glycemic variability indexes would be better predictors of MACE. Using continuous glucose measurement for 48 h, it has been shown that significant glycemic variability is a more powerful predictor of MACE at 1 year than admission glycemia The measurement of glycemic variability is mainly possible thanks to the development of CGM (continuous glucose measurement).

To our knowledge, no study has been interested in evaluating the predictive value of the various glycemic parameters measured by CGM.

Published studies have used continuous glucose measurements for very short periods (24 or 72 hours maximum), which limits these measurements.

The freestyle libre Pro iQ (FSLPro iQ) is a professional sensor for continuous, non-invasive interstitial glucose measurement allowing the recording of glycemic parameters for 2 weeks.

Our hypothesis is that glycaemic parameters, alone or in combination with each other or with other patient risk factors, measured with the Freestyle libre Pro iQ have a significant prognostic value in terms of cardiovascular clinical events at 12 months in a population of patients with ACS managed as standard and followed up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ACS managed in a cardiac intensive care unit (ICU). The diagnosis of ACS will be made in the presence of chest pain with ST-segment elevation on the ECG for STEMI or ST-segment change and/or a positive troponin cycle (values in accordance with the center's protocol) for NSTEMI.

Exclusion Criteria:

* Subjects in cardiogenic or septic shock
* Subjects with ACS initially managed in a non-investigating center
* Failure to obtain free, informed, written consent signed by the participant and investigator upon admission to the ICU
* Person participating in another research study with an ongoing exclusion period
* Subjects participating in a study that may have an impact on post ACS prognosis
* Person deprived of his or her rights, person under guardianship or curatorship
* Person deprived of liberty (by judicial or administrative decision)
* Persons whose physical and/or psychological health is severely impaired, which, in the opinion of the investigator, may affect the participant's compliance to the study
* Pregnant or breastfeeding women
* Person who is not affiliated to a social security system or who is a beneficiary of such a system.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 850 (Estimated)
Dates: Start 2023-11-06 (Actual); Primary Completion 2028-05-06 (Estimated); Study Completion 2028-05-06 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular events | 12 months
  Occurrence within 12 months of hospital discharge of a composite end point including cardiovascular clinical events: recurrent MI, cardiovascular death, stroke, rhythm disturbance, and/or heart failure requiring hospitalization.

SECONDARY OUTCOMES:
Diabetes | 12 months
  Incidence of diabetes at 12 months in nondiabetic subjects admitted for ACS: measurement of fasting venous glucose (≥ 1.26g/l) and HbA1c (≥ 6.5%).
Diabetes | 2 months
  Incidence of diabetes at 1-2 months in nondiabetic subjects admitted for ACS: fasting venous glucose measurement (≥ 1.26g/L) and HbA1c (≥ 6.5%).

CONTACTS AND LOCATIONS:
Locations (9):
- France (9):
  - Hospital of Béziers, Béziers
  - University Hospital of Bordeaux, Bordeaux
  - University Hospital of Montpellier, Montpellier
  - University Hospital of Nîmes, Nîmes
  - AP-HP Lariboisière Hospital, Paris
  - APHP - Hôpital Européen Georges Pompidou, Paris
  - Hospital of Pau, Pau
  - University Hospital of Toulouse, Toulouse
  - Vannes Bretagne Atlantique Hospital, Vannes